CLINICAL TRIAL: NCT06449534
Title: The Effect of the Treatment Environment on Pain, Function, Self Efficacy and Satisfaction in Rotator Cuff Related Shoulder Pain
Brief Title: The Effect of the Treatment Environment on Pain, Function, Self Efficacy and Satisfaction in RCRSP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Merve Koyuncu Cenikli, Research Asistant, PT, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2150060
Record Dates: First submitted 2024-05-27; First posted 2024-06-10 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Shoulder Pain; Subacromial Pain Syndrome; Rotator Cuff Syndrome of Shoulder and Allied Disorders
Keywords: Therapeutic Environment; Contextual Factors; Exercise Therapy
MeSH Terms: conditions — Shoulder Pain | interventions — Patient Education as Topic; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The enriched therapeutic environment group (Group 1) (Experimental): Group 1 will receive treatment in a physiotherapy unit which has following characteristics ; enlightened with sunlight, has a view of green trees and includes other participants exercising. Patients will receive a treatment consisting of patient education, exercise therapy and cold application for a total of 15 sessions, 3 times a week. Each session will last approximately 60 minutes. After the patient education and exercise therapy is completed, the participants will listen to classical music pieces selected by us during 15 minutes of cold application.
  Interventions: Behavioral: Patient Education; Behavioral: Exercise Therapy; Behavioral: Cold Application
- The isolated therapeutic environment group (Group 2). (Experimental): Group 2 will receive treatment in a quiet single room. The room is illuminated by artificial light, curtains are closed so that patients cannot see outside view. Patients will receive a treatment consisting of patient education, exercise therapy and cold application for a total of 15 sessions, 3 times a week. Each session will last approximately 60 minutes. After the patient education and exercise therapy is completed, the participants will rest silently for 15 minutes of cold application.
  Interventions: Behavioral: Patient Education; Behavioral: Exercise Therapy; Behavioral: Cold Application

INTERVENTIONS:
Behavioral: Patient Education — It includes evaluation of the treatment process and past sessions. Simple shoulder biomechanics, function, and what caused the injury were explained to the patients. In order to increase patients' participation in treatment, it was emphasized what the treatment does and that the patient should cooperate in order to heal. During their treatment, patients are instructed to regulate their daily living activities, avoid overhead and repetitive movements of the arm, bags weighing more than 2-3 kg, etc. It was recommended not to carry them. Patients were informed about alternative sleeping positions.
Behavioral: Exercise Therapy — Participants in both groups were included in a structured exercise program consisting of exercises recommended in the literature. This exercise program includes joint range of motion exercises, stretching exercises and strengthening exercises and was carried out under the supervision of a physiotherapist for 6 weeks. Joint range of motion and strengthening exercises are recommended as 3 sets of 10 repetitions, and stretching exercises are recommended as 5 repetitions for 20 seconds. Exercises appropriate to the patients' clinical conditions and progression were selected by the physiotherapist and included in the program.
Behavioral: Cold Application — Following each exercise treatment, cold-pack will be applied for 15 minutes. During col-pack application, patients in the Group 1 group will listen to classical music selected by us, while patients in the Group 2 will rest quietly. There are a total of 40 songs by Bach, Mozart, Beethoven and Andre Rieu on our CD player, and patients have the right to choose and listen to the song they want.

SUMMARY:
Brief Summary

The aim of this randomized controlled study is to reveal the short-term effects of physical and social factors in different therapeutic environments on patients with rotator cuff related shoulder pain following the same exercise program. The main questions it aims answer are:

* Is there any difference in terms of pain levels among groups with rotator cuff related shoulder pain who treated in different therapeutic settings.
* Is there any difference in terms of functionality and self-efficacy among groups with rotator cuff related shoulder pain who treated in different therapeutic settings.

DETAILED DESCRIPTION:
The investigators will include patients who applied to the physiotherapy clinic of Kadikoy Florence Nightingale Medical Center with the complaint of shoulder pain. 46 individuals who volunteer to participate in the study will be included. Participants will be randomised through a computer-based randomization program into two groups; the enriched therapeutic environment group (Group 1) and the isolated therapeutic environment group (Group 2). The same treatment including patient education, exercise therapy and ice application will be performed to both groups. Participants will receive a total of 15 sessions of treatment, 3 sessions per week. Before the treatment, 3rd week, 6th week and 12th week, the following evaluations will be made to both groups; Numerical Pain Rating Scale (NPRS) to asses pain, Arm, Shoulder, Hand Problems Quick Survey (Quick-DASH) and Western Ontario Rotator Cuff Index (WORC) to asses functionality, Pain Self-Efficacy Questionnaire (PSEQ) to asses self efficacy and Global Scale of Change (GRC) to asses the effectiveness of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* diagnosed with impingement syndrome, subacromial bursitis, rotator cuff tendinopathy or partial rotator cuff tear
* pain level between 3-7 according to visual analog scale
* pain persisted for at least 3 months

Exclusion Criteria:

* having a full-thickness or massive rotator cuff tear
* history of shoulder surgery
* having a musculoskeletal disease that prevents exercise
* having a neurological disease or psychological disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Baseline, 3rd week, 6th week
  Participants' pain at rest, at night and during activity was measured using the NPRS. The NPRS is an 11-point scale that can be scored from 0 to 10. A score of zero (0) indicates "no pain" and 10 indicates score defines "the most severe pain". The patient will be asked to mark shoulder pain on the scale

SECONDARY OUTCOMES:
Quick - The Disabilities of the Arm, Shoulder and Hand (Quick DASH) Questionnaire | Baseline, 3rd week, 6th week, 12th week
  Q-DASH is a questionnaire developed to assess upper extremity functioning and symptoms based on self-report of patients. The total score of the scale ranges from 0-100 points and similar to SPADI, a high score is considered as high functional disability.
Western Ontario Rotator Cuff (WORC) Index | Baseline, 3rd week, 6th week, 12th week
  WORC is a functional test which consists of 5 sections and a total of 21 questions assessing the physical symptoms, sports/leisure time activities, work, lifestyle, emotions that are affected by the shoulder problem. Each question is rated on a scale of 0-100 mm. Patients are scored between 0 and 2100 in total, with 2100 being the worst score.
Pain Self-Efficacy Questionnaire (PSEQ) | Baseline, 3rd week, 6th week, 12th week
  The Pain and Self-Efficacy questionnaire consists of 10 questions and it assesses multiple domains of self-efficacy related to social and physical functioning. Each item is rated on a 7-point Likert-type scale (0: I am not at all confident, 6: I am completely confident). The total score ranges from 0 to 60, with higher scores indicating greater self-efficacy for functioning despite pain.
Global Rating of Change, GRC | Baseline, 3rd week, 6th week, 12th week
  The Global Rating of Change (GRC) is specifically designed to determine the impact of an intervention in musculoskeletal problems, to chart the clinical course of a condition and to measure a patient's improvement or deterioration over time. When using the GRC scale, the patient being assessed must have a certain cognitive level because the patient's ability to recall and measure the pre-treatment state is required. In our study, a scale consisting of 5 levels will be used (-2: much worse, -1: worse, 0: same, 1: better, 2: much better).

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul University Cerrahpasa Faculty of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No